CLINICAL TRIAL: NCT05282004
Title: An Open-label, Single-arm, Multicenter Study in Patients With Neovascular Age-related Macular Degeneration to Evaluate the Safety of SOK583A1 (40 mg/mL), a Proposed Aflibercept Biosimilar Product, Provided in a Vial Kit
Brief Title: Study of the Safety of Use of Intravitreal SOK583A1 Provided in a Vial Kit
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSOK583A12303
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Results first posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-04

CONDITIONS: Neovascular Age-related Macular Degeneration (nAMD)
Keywords: Open label study,; intravitreal injection,; biosimilar,; aflibercept,; vial kit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SOK583A1 (Experimental): SOK583A1 will be provided in a vial kit, with 40 mg/mL of aflibercept solution for IVT injection (2 mg/0.05 mL)
  Interventions: Drug: SOK583A1

INTERVENTIONS:
Drug: SOK583A1 — SOK583A1 will be provided in a vial kit, with 40 mg/mL of aflibercept solution for IVT injection (2 mg/0.05 mL)

SUMMARY:
This is a single-arm, open-label study where all patients will receive a single injection of SOK583A1 (40 mg/mL) provided in a vial kit at Baseline. The total study duration for the individual participant is approximately 31 days.

DETAILED DESCRIPTION:
Subjects with nAMD received a single dose of study treatment (2 mg SOK583 in 0.05 mL) in line with the Eylea USPI, which recommends a dose of 2 mg aflibercept (0.05 mL) administered by IVT injection. Only subjects already under IVT Eylea treatment and hence familiar with the IVT procedure were eligible for the study. Administration of the study treatment was embedded into their routine treatment scheme.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 50 years of age at baseline
* Patients diagnosed with nAMD (uni- or bilateral)
* Patients already under IVT Eylea treatment (last injection of the induction period or maintenance phase)
* Willing and able to comply with all study procedures, and be likely to complete the study
* Signed informed consent must be obtained before any assessment is performed

Exclusion Criteria:

* Active, suspected or recent (within 4 weeks) intraocular inflammation (grade trace or above) in the study eye at baseline, which is of clinical significance according to the investigator's judgment, such as active infections of the anterior segment; this includes conjunctivitis (except mild blepharitis), keratitis, scleritis, idiopathic or autoimmune associated uveitis or endophthalmitis
* Any uncontrolled ocular hypertension or glaucoma in the study eye (defined as IOP ≥ 26 mmHg, despite treatment with anti-glaucomatous medication)
* History of a medical, ocular or non-ocular condition, that in the judgment of the investigator, would preclude a safe administration of investigational product
* Visual acuity Score (VAS) worse than 20/200 on a Snellen chart, the generally accepted level of legal blindness
* Topical ocular corticosteroids administered for at least 30 consecutive days within 3 months prior to screening
* Systemic treatment with long-acting corticosteroids (more than 10 mg prednisolone equivalent) within 3 months prior to screening Current or planned use of systemic medications known to be toxic to the lens, retina or optic nerve, including deferoxamine, chloroquine/hydroxychloroquine, tamoxifen, phenothiazines and ethambutol
* Any invasive intraocular surgery, prior long-acting therapeutic agent, or ocular drug release device implantation (approved or investigational) in the study eye any time during the past 3 months
* Receipt of any systemic anti-VEGF within the last 6 months prior to enrollment
* Uncontrolled hypertension (defined as a systolic value ≥ 160 mmHg or diastolic value ≥ 100 mmHg at Screening)
* Participants who do not comply with the local COVID-19 regulations of the study site

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Sandoz Investigational Site, Poway, California
  - Sandoz Investigational Site, Marietta, Georgia
  - Sandoz Investigational Site, Oak Forest, Illinois
  - Sandoz Investigational Site, Liverpool, New York
  - Sandoz Investigational Site, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 5 study sites in the USA.
Groups:
- SOK583A1 40 mg/mL: SOK583A1 was provided in a vial kit, with 40 mg/mL of aflibercept solution for IVT injection (2 mg/0.05 mL)
Period: Overall Study
Arm/Group | SOK583A1 40 mg/mL
Started | 36
Completed | 34
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | SOK583A1 40 mg/mL
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.9 (8.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 36
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Ocular Treatment Emergent Adverse Events
Description: Number of participants with ocular treatment emergent adverse events were reported.
Time Frame: 31 days
Population: Full analysis set (FAS): FAS included all participants who received an injection of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | SOK583A1 40 mg/mL
Number analyzed (Participants) | 36
Participants | 16

2. Primary Outcome: Number of Participants With Non-ocular Treatment Emergent Adverse Events
Description: Number of participants with non-ocular treatment emergent adverse events were reported.
Time Frame: 31 days
Population: Full analysis set (FAS): FAS included all participants who received an injection of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | SOK583A1 40 mg/mL
Number analyzed (Participants) | 36
Participants | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study for 31 days
Description: Any signs or symptoms were collected throughout the study for 31 days
Arm/Group | SOK583A1 40 mg/mL
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 2/36
Other Adverse Events (participants affected / at risk) | 17/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOK583A1 40 mg/mL (N=36)
Cystitis (Infections and infestations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOK583A1 40 mg/mL (N=36)
Conjunctival haemorrhage (Eye disorders) | 2
Vitreous floaters (Eye disorders) | 1
COVID-19 (Infections and infestations) | 1
Intraocular pressure increased (Investigations) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Sandoz' agreements with its investigators may vary. However, Sandoz does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT05282004/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT05282004/SAP_001.pdf